CLINICAL TRIAL: NCT00247702
Title: Study of the Association of Warfarin Dosage and Plasma Enantiomer Concentration With the Gene Polymorphisms of CYP and VKOR
Brief Title: The Association of Warfarin Dosage and Plasma Enantiomer Concentration With the Gene Polymorphisms of CYP and VKOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 940609
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2005-11-02 (Estimated); Status verified 2005-07

CONDITIONS: Deep Venous Thromboembolism
Keywords: CYP2C9; VKORC1; polymorphism; warfarin
MeSH Terms: conditions — Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2 | interventions — Warfarin

INTERVENTIONS:
Drug: warfarin

SUMMARY:
Oral warfarin anticogulation for the prevention and treatment of patients with venous thromboembolism is one of the most used therapies in clinical practice. Patients require different dosage to achieve the target therapeutic anticoagulation. Optimal dosage and bleeding complication are two most clinical concerns. Besides of multiple individual factors (e.g. age, dietary intake, vitamin supplement, drug compliance etc.), some genetic factors may determine the drug requirement and safety.

The cytochrome P450 CYP2C9 is a liver enzyme required for the oxidative metabolism of warfarin. The vitamin K epoxide redutase (VKOR) is a liver enzyme associated with the reuse of the oxidative hydroquinone form of vitamin K. The VKOR enzyme is the target of warfarin. Recent studies revealed both genes may determine the pharmacodynamic of warfarin anticogualation. To date, there are more than thirteen identified polymorphism at CYP2C9 gene. Majority of those variant polymorphisms may decrease the warfarin requirement. The VKOR complex subunit 1 (VKORC1) is a newly identified gene. Some polymorphisms also were reported.

As we know, the Chinese patients need a lower dosage of warfarin in comparison with the Caucasian patients. We are interested in finding the genetic causes of Taiwneses Chinese patients. In our study we will first identify the polymorphism patterns of these two genes in normal population. Then, we will try to find the association between these polymorphism and patient warfarin requirement. Our pharmacogenetics study will be valuable for prevention of bleeding complication of warfarin treatment in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Use warfarin therapy for at least two months before study
* Stable INR value during recent three months

Exclusion Criteria:

* higher age(>80 y/o)
* liver and renal dysfunction
* alcohol abuse
* BMI<18kg/m2
* coadministered medicine that can affect pharmacokinetics or pharmacodynamics of warfarin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Tasy Wei, Doctor, Study Chair — National Taiwan Univerisity Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan